CLINICAL TRIAL: NCT04336696
Title: Is Routine Dissection of Central Lymph Node Necessary for Papillary Thyroid Carcinoma, T1-2 N0?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bassem Mohamed Sieda (Other Government)
Responsible Party: Sponsor-Investigator, Bassem Mohamed Sieda, Assistant Professor of general surgery, Faculty of medicine, Zagazig University
Organization: Zagazig University (Other Government)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 0000-0002-9836-9580
Record Dates: First submitted 2020-04-01; First posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Papillary Thyroid Carcinoma
Keywords: papillary carcinoma; recurrence of PTC; Radio-iodine therapy for PTC
MeSH Terms: conditions — Thyroid Cancer, Papillary; Carcinoma, Papillary

STUDY DESIGN:
Intervention Model Description: prospective cohort study
Who Masked: Participant, Investigator
Masking Description: guuartor of study, only participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Comparison between the studied groups regarding management. (Active Comparator): The postoperative RAI scan after 1 month, showed a positive residual tumour in lateral LN in 70 patients in the controlled group and 13 patients in Group II, 8 patients in group III. In group I, Patients with residuals were submitted to RAI ablation.
  Interventions: Procedure: Total thyroidectomy and central neck dissection
- Recurrence free survival (Other): patients with total thyroidectomy only had shorter recurrence free survival
  Interventions: Procedure: Total thyroidectomy and central neck dissection

INTERVENTIONS:
Procedure: Total thyroidectomy and central neck dissection

SUMMARY:
study assigned into three groups, Group I was the control group operated by total thyroidectomy and retrospectively followed, where the other two groups Operated by Total thyroidectomy and central neck dissection. Recurrence Free Survival (RFS) was the main issue of the study and calculated as the time from date of surgery to date of relapse or the most recent follow-up contact that patient was known as relapse-free, Study exclusively studied the outcome and advantage of central neck dissection

DETAILED DESCRIPTION:
informed consent taken, study was a prospective cohort study, with controlled group a retrospectively. patients ablated by total thyroidectomy only who failed to achieve ablation with the first dose of iodine 131I may be dynamically risk stratified as high-risk category and managed aggressively. N0 patients will benefit and ablated by total thyroidectomy and prophylactic central neck dissection, PCND decreases the residual, increase the RFS and patients without residual do not need adjuvant RAI therapy except in high risk group. Histological grading, size of the primary tumour, the extension of PTC, the extent of surgery were found to be a strong predicting factor for recurrence-free survival

Locoregional recurrence cases always found more in male patients aged more than 45 years old. Size of the primary tumour and the extent of surgery was a significant factor for RFS,

ELIGIBILITY:
Inclusion Criteria:

* Age ≥20 years, Histopathology proved PTC, with no lymph nodes detected (N0)

Exclusion Criteria:

* Younger age ≤20 years. Prior thyroidectomy, previous radiation exposure, postoperative radioactive iodine therapy, Histopathology report of any type of malignancy other than PTC or patients did not complete their postoperative follow-up period. PTC With N1 or N2

Ages: 42 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 199 (Estimated)
Dates: Start 2016-11-02 (Actual); Primary Completion 2020-04-03 (Estimated); Study Completion 2020-05-03 (Estimated)

PRIMARY OUTCOMES:
recurrence free survival | 21 months
  recurrence free survival calculated from first day of diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University Hospitals, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Yes
after aprovel, recommendation of study will be shared with other researchers
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year

REFERENCES:
- [Result] Viola D, Materazzi G, Valerio L, Molinaro E, Agate L, Faviana P, Seccia V, Sensi E, Romei C, Piaggi P, Torregrossa L, Sellari-Franceschini S, Basolo F, Vitti P, Elisei R, Miccoli P. Prophylactic central compartment lymph node dissection in papillary thyroid carcinoma: clinical implications derived from the first prospective randomized controlled single institution study. J Clin Endocrinol Metab. 2015 Apr;100(4):1316-24. doi: 10.1210/jc.2014-3825. Epub 2015 Jan 15. PMID 25590215
- [Result] Kim K, Kim JH, Park IS, Rho YS, Kwon GH, Lee DJ. The Updated AJCC/TNM Staging System for Papillary Thyroid Cancer (8th Edition): From the Perspective of Genomic Analysis. World J Surg. 2018 Nov;42(11):3624-3631. doi: 10.1007/s00268-018-4662-2. PMID 29750323